CLINICAL TRIAL: NCT02064192
Title: Comparative Effectiveness Research to Assess the Use of Primary ProphylacTic Implantable Cardioverter Defibrillators in Europe
Acronym: EU-CERT-ICD
Status: Completed | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Markus Zabel, Associate Professor of Medicine, University Medical Center Goettingen
Other Study IDs: EU 602299
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Coronary Artery Disease; Myocardial Infarction; Dilated Cardiomyopathy; Implantable Defibrillator User
Keywords: defibrillator, implantable cardioverter; sudden cardiac death; primary prophylaxis; risk stratification
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Cardiomyopathy, Dilated; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood sample for genetic analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ICD Group (n=1500): First ICD device implantation (after baseline assessments) is not part of this observational study and is carried out in the responsibility of the treating physician, all ICD-devices will undergo unique standard programming to ensure comparability of ICD shock events between patients.
- Control Group (n=750): Patients who fulfill inclusion criteria but do not receive an ICD device will be followed as part of the Control Group

SUMMARY:
The "EUropean Comparative Effectiveness Research to assess the use of primary prophylacTic Implantable Cardioverter Defibrillators (EU-CERT-ICD)" is a modular research project to study the effectiveness of prophylactic ICDs in a prospective study, a retrospective registry, and meta-analyses of existing evidence on the subject.

DETAILED DESCRIPTION:
The prospective study part is an observational, prospective multi-centre study which aims to enrol 2500 patients with ischemic or dilated cardiomyopathy and primary prophylactic ICD indication for reduced left ventricular ejection fraction (LVEF) according to current guidelines. According to the treating physician's decision and preference which is independent from study participation, patients are recruited into one of two groups: patients directly prior to first ICD implantation (ICD Group), or patients who are not considered for prophylactic ICD treatment by the physician or are considered but refuse ICD treatment (Control Group). Patients will undergo simple 12-lead electrocardiogram (ECG) and Holter ECG diagnostics at baseline as well as genetic biobanking at entry to the study. All patients will be subsequently followed for at least 1 year and up to 4 years. Co-primary endpoints are all-cause mortality and appropriate ICD shocks.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or dilated cardiomyopathy and recommendation for primary prophylactic ICD treatment following current international treatment guidelines
* Written informed consent
* If ICD implantation is planned, enrollment and study baseline testing needs to be completed before de-novo ICD implantation

Exclusion Criteria:

* Permanent atrial fibrillation or atrial fibrillation at baseline in case more than 15% of such patients at a given time have been enrolled
* Indication for secondary prophylactic ICD treatment
* Indication or candidate for cardiac resynchronization therapy
* AV block II°-III° at resting heart rates
* Implanted pacemaker
* Unstable cardiac disease such as decompensated heart failure (NYHA functional class IV) or acute coronary syndrome
* Participation in other clinical trials which exclude enrolment in other trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are eligible for primary prophylactic ICD implantation and potentially eligible for study participation will be identified based on echocardiographic and/or 12 lead ECG results. For ICD Group patients, screening will be shortly before scheduled ICD implantation. For Control Group patients, the time span between primary diagnosis of eligibility for primary ICD implantation and the date of the primary diagnosis of cardiomyopathy must be recorded in the eCRF, together with how and when the decision not to prescribe a defibrillator was reached. Control group will be recruited from patients with ischemic or dilated cardiomyopathies and LVEF ≤ 35%. Patients scheduled for ICD implantation (ICD Group) undergo screening and baseline assessments prior to ICD implantation. Patients for the Control Group will undergo baseline assessments as soon as possible after screening. Baseline assessments are identical for the ICD Group and the Control Group.
Sampling Method: Probability Sample
Enrollment: 2285 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
All-Cause Mortality | one to five years
  Co-Primary Endpoint
First Appropriate ICD Shock | one to five years
  Co-Primary Endpoint

SECONDARY OUTCOMES:
Time to First Inappropriate Shock | one to five years
Sudden Cardiac Death | one to five years
Cardiac Death | one to five years
Non-Cardiac Death | one to five years
Arrhythmogenic Syncope | one to five years
  presumed arrhythmogenic syncopes (per the judgment of each investigator and the endpoint committee)
Resuscitation | one to five years
  successful resuscitation for ventricular tachyarrhythmias (especially in the non ICD Control Group)
Any ICD Shock | one to five years
  any ICD shock (appropriate or inappropriate)
Atrial Fibrillation | one to five years
  atrial fibrillation (if documented), defined as an atrial tachyarrhythmia >250 beats per minute (bpm) lasting at least 30 seconds is considered as secondary endpoint
Quality of Life | one to five years
  Quality of life (QoL) will be assessed using the questionnaires SF 36, MacNew and Florida Patient Acceptance Survey
Device Revision / Device Replacement | one to five years
  the secondary endpoint Device Revision/Replacement will be recorded as electrode dislocation/revision, device revision for pocket hematoma, perforation, or infection, device exchange due to malfunction, battery exhaustion, other reason, or upgrade to dual chamber or CRT-D
Costs and Cost-Effectiveness | one to five years
  the secondary endpoint "Costs" will be assessed using patient questionnaires to the German-speaking study sites, an extension to other participating countries will be decided during the study, the assessment of cost-effectiveness will be realised by comparing cost-results with regard to changes in QoL

CONTACTS AND LOCATIONS:
Overall Officials: Markus Zabel, MD, Principal Investigator — University Medical Center Goettingen
Locations (42):
- KU Leuven, Div. of Cardiology, Leuven, Belgium
- Bulgaria (4):
  - National Heart Hospital, Dept. of Cardiology, Sofia
  - Acibadem City Clinic Tokuda Hospital, Div. of Cardiology, Sofia
  - St. Ekaterina Hospital, Div. of Cardiology, Sofia
  - St. Anna University Hospital for Active Treatment, Div. of Cardiology, Sofia
- Croatia (5):
  - Magdalena Clinic, Krapinske Toplice
  - Klinički bolnički centar Rijeka, Div. of Cardiology, Rijeka
  - Klinički bolnički centar Split, Div. of Cardiology, Split
  - Opća Bolnica Zadar, Div. of Cardiology, Zadar
  - Klinički bolnički centar Sestre milosrdnice, Div. of Cardiology, Zagreb
- Czechia (2):
  - Masaryk University Hospital Brno, Div. of Cardiology, Brno
  - Palacky University Hospital Olomouc, Div. of Cardiology, Olomouc
- Denmark (2):
  - Rigshospitalet, Div. of Cardiology, Copenhagen
  - Gentofte Hospital, Div. of Cardiology, Hellerup
- Department of Internal Medicine, University of Oulu, Oulu, Finland
- Germany (14):
  - CharitéCentrum 1 Health and Human Sciences, Institute for Social Medicine, Epidemiology and Health Economics, Berlin
  - Charitè Virchow Klinikum (CVK), Div. of Cardiology, Berlin
  - Vivantes Humboldt Klinikum, Div. of Cardiology, Berlin
  - St. Marien-Hospital, Div. of Cardiology, Bonn
  - Klinikum Reinkenheide, Div. of Cardiology, Bremerhaven
  - University Medical Center, Div. of Cardiology, Göttingen
  - Asklepios Klinikum Barmbek, Div. of Cardiology, Hamburg
  - Herz im Zentrum, Hanover
  - Klinikum Ludwigsburg, Div. of Cardiology, Ludwigsburg
  - Department of Cardiovascular Diseases, German Heart Centre Munich, Technische Universität München, Munich
  - Ludwig-Maximilians-University, Div. of Cardiology, Munich
  - University Hospital Regensburg, Div. of Cardiology, Regensburg
  - University Hospital Tuebingen, Div. of Cardiology, Tübingen
  - Klinikum Weiden, Div. of Cardiology, Weiden
- Attikon University Hospital, Div. of Cardiology, Athens, Greece
- Semmelweis University Heart and Vascular Center, Budapest, Hungary
- Universitair Medisch Centrum Utrecht, Dept. of Physiology & Cardiology, Utrecht, Netherlands
- Poland (3):
  - Medical University of Lodz, Lodz
  - Heliodor Swiecicki University Hospital, Div. of Cardiology, Poznan
  - Cardinal Stefan Wyszynski Institute of Cardiology (IKARD), Warsaw
- Slovakia (2):
  - Stredoslovenský ústav srdcových a cievnych chorôb (SUSSCH), Banská Bystrica
  - Slovak Medical University, Heart Center, Bratislava
- Hospital Clínic, Universitat de Barcelona, Barcelona, Spain
- Sweden (2):
  - Skane University Hospital, Div. of Cardiology, Lund
  - Karolinska Institute, Div. of Cardiology, Stockholm
- University Hospital Basel, Div. of Cardiology, Basel, Switzerland
- St. Paul's Cardiac Electrophysiology, London, Purley, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hlatky MA, Douglas PS, Cook NL, Wells B, Benjamin EJ, Dickersin K, Goff DC, Hirsch AT, Hylek EM, Peterson ED, Roger VL, Selby JV, Udelson JE, Lauer MS. Future directions for cardiovascular disease comparative effectiveness research: report of a workshop sponsored by the National Heart, Lung, and Blood Institute. J Am Coll Cardiol. 2012 Aug 14;60(7):569-80. doi: 10.1016/j.jacc.2011.12.057. Epub 2012 Jul 11. PMID 22796257
- [Background] Huikuri HV, Castellanos A, Myerburg RJ. Sudden death due to cardiac arrhythmias. N Engl J Med. 2001 Nov 15;345(20):1473-82. doi: 10.1056/NEJMra000650. No abstract available. PMID 11794197
- [Background] Bardy GH, Lee KL, Mark DB, Poole JE, Packer DL, Boineau R, Domanski M, Troutman C, Anderson J, Johnson G, McNulty SE, Clapp-Channing N, Davidson-Ray LD, Fraulo ES, Fishbein DP, Luceri RM, Ip JH; Sudden Cardiac Death in Heart Failure Trial (SCD-HeFT) Investigators. Amiodarone or an implantable cardioverter-defibrillator for congestive heart failure. N Engl J Med. 2005 Jan 20;352(3):225-37. doi: 10.1056/NEJMoa043399. PMID 15659722
- [Background] Koller MT, Schaer B, Wolbers M, Sticherling C, Bucher HC, Osswald S. Death without prior appropriate implantable cardioverter-defibrillator therapy: a competing risk study. Circulation. 2008 Apr 15;117(15):1918-26. doi: 10.1161/CIRCULATIONAHA.107.742155. Epub 2008 Apr 7. PMID 18391108
- [Background] Tung R, Zimetbaum P, Josephson ME. A critical appraisal of implantable cardioverter-defibrillator therapy for the prevention of sudden cardiac death. J Am Coll Cardiol. 2008 Sep 30;52(14):1111-21. doi: 10.1016/j.jacc.2008.05.058. PMID 18804736
- [Background] Moss AJ, Schuger C, Beck CA, Brown MW, Cannom DS, Daubert JP, Estes NA 3rd, Greenberg H, Hall WJ, Huang DT, Kautzner J, Klein H, McNitt S, Olshansky B, Shoda M, Wilber D, Zareba W; MADIT-RIT Trial Investigators. Reduction in inappropriate therapy and mortality through ICD programming. N Engl J Med. 2012 Dec 13;367(24):2275-83. doi: 10.1056/NEJMoa1211107. Epub 2012 Nov 6. PMID 23131066
- [Background] MacFadden DR, Crystal E, Krahn AD, Mangat I, Healey JS, Dorian P, Birnie D, Simpson CS, Khaykin Y, Pinter A, Nanthakumar K, Calzavara AJ, Austin PC, Tu JV, Lee DS. Sex differences in implantable cardioverter-defibrillator outcomes: findings from a prospective defibrillator database. Ann Intern Med. 2012 Feb 7;156(3):195-203. doi: 10.7326/0003-4819-156-3-201202070-00007. PMID 22312139
- [Background] Cowie MR, Marshall D, Drummond M, Ferko N, Maschio M, Ekman M, de Roy L, Heidbuchel H, Verboven Y, Braunschweig F, Linde C, Boriani G. Lifetime cost-effectiveness of prophylactic implantation of a cardioverter defibrillator in patients with reduced left ventricular systolic function: results of Markov modelling in a European population. Europace. 2009 Jun;11(6):716-26. doi: 10.1093/europace/eup068. Epub 2009 Apr 9. PMID 19359333
- [Background] Kramer DB, Friedman PA, Kallinen LM, Morrison TB, Crusan DJ, Hodge DO, Reynolds MR, Hauser RG. Development and validation of a risk score to predict early mortality in recipients of implantable cardioverter-defibrillators. Heart Rhythm. 2012 Jan;9(1):42-6. doi: 10.1016/j.hrthm.2011.08.031. Epub 2011 Sep 3. PMID 21893137
- [Background] Al-Khatib SM, Hellkamp A, Bardy GH, Hammill S, Hall WJ, Mark DB, Anstrom KJ, Curtis J, Al-Khalidi H, Curtis LH, Heidenreich P, Peterson ED, Sanders G, Clapp-Channing N, Lee KL, Moss AJ. Survival of patients receiving a primary prevention implantable cardioverter-defibrillator in clinical practice vs clinical trials. JAMA. 2013 Jan 2;309(1):55-62. doi: 10.1001/jama.2012.157182. PMID 23280225
- [Background] Schmidt G, Malik M, Barthel P, Schneider R, Ulm K, Rolnitzky L, Camm AJ, Bigger JT Jr, Schomig A. Heart-rate turbulence after ventricular premature beats as a predictor of mortality after acute myocardial infarction. Lancet. 1999 Apr 24;353(9162):1390-6. doi: 10.1016/S0140-6736(98)08428-1. PMID 10227219
- [Background] Bauer A, Kantelhardt JW, Barthel P, Schneider R, Makikallio T, Ulm K, Hnatkova K, Schomig A, Huikuri H, Bunde A, Malik M, Schmidt G. Deceleration capacity of heart rate as a predictor of mortality after myocardial infarction: cohort study. Lancet. 2006 May 20;367(9523):1674-81. doi: 10.1016/S0140-6736(06)68735-7. PMID 16714188
- [Background] Zabel M, Malik M, Hnatkova K, Papademetriou V, Pittaras A, Fletcher RD, Franz MR. Analysis of T-wave morphology from the 12-lead electrocardiogram for prediction of long-term prognosis in male US veterans. Circulation. 2002 Mar 5;105(9):1066-70. doi: 10.1161/hc0902.104598. PMID 11877356
- [Background] Thomsen MB, Volders PG, Beekman JD, Matz J, Vos MA. Beat-to-Beat variability of repolarization determines proarrhythmic outcome in dogs susceptible to drug-induced torsades de pointes. J Am Coll Cardiol. 2006 Sep 19;48(6):1268-76. doi: 10.1016/j.jacc.2006.05.048. Epub 2006 Aug 28. PMID 16979017
- [Background] Exner DV, Kavanagh KM, Slawnych MP, Mitchell LB, Ramadan D, Aggarwal SG, Noullett C, Van Schaik A, Mitchell RT, Shibata MA, Gulamhussein S, McMeekin J, Tymchak W, Schnell G, Gillis AM, Sheldon RS, Fick GH, Duff HJ; REFINE Investigators. Noninvasive risk assessment early after a myocardial infarction the REFINE study. J Am Coll Cardiol. 2007 Dec 11;50(24):2275-84. doi: 10.1016/j.jacc.2007.08.042. Epub 2007 Nov 26. PMID 18068035
- [Background] Ellinor PT, Lunetta KL, Albert CM, Glazer NL, Ritchie MD, Smith AV, Arking DE, Muller-Nurasyid M, Krijthe BP, Lubitz SA, Bis JC, Chung MK, Dorr M, Ozaki K, Roberts JD, Smith JG, Pfeufer A, Sinner MF, Lohman K, Ding J, Smith NL, Smith JD, Rienstra M, Rice KM, Van Wagoner DR, Magnani JW, Wakili R, Clauss S, Rotter JI, Steinbeck G, Launer LJ, Davies RW, Borkovich M, Harris TB, Lin H, Volker U, Volzke H, Milan DJ, Hofman A, Boerwinkle E, Chen LY, Soliman EZ, Voight BF, Li G, Chakravarti A, Kubo M, Tedrow UB, Rose LM, Ridker PM, Conen D, Tsunoda T, Furukawa T, Sotoodehnia N, Xu S, Kamatani N, Levy D, Nakamura Y, Parvez B, Mahida S, Furie KL, Rosand J, Muhammad R, Psaty BM, Meitinger T, Perz S, Wichmann HE, Witteman JC, Kao WH, Kathiresan S, Roden DM, Uitterlinden AG, Rivadeneira F, McKnight B, Sjogren M, Newman AB, Liu Y, Gollob MH, Melander O, Tanaka T, Stricker BH, Felix SB, Alonso A, Darbar D, Barnard J, Chasman DI, Heckbert SR, Benjamin EJ, Gudnason V, Kaab S. Meta-analysis identifies six new susceptibility loci for atrial fibrillation. Nat Genet. 2012 Apr 29;44(6):670-5. doi: 10.1038/ng.2261. PMID 22544366
- [Background] Seegers J, Vos MA, Flevari P, Willems R, Sohns C, Vollmann D, Luthje L, Kremastinos DT, Flore V, Meine M, Tuinenburg A, Myles RC, Simon D, Brockmoller J, Friede T, Hasenfuss G, Lehnart SE, Zabel M; EUTrigTreat Clinical Study Investigators. Rationale, objectives, and design of the EUTrigTreat clinical study: a prospective observational study for arrhythmia risk stratification and assessment of interrelationships among repolarization markers and genotype. Europace. 2012 Mar;14(3):416-22. doi: 10.1093/europace/eur352. Epub 2011 Nov 23. PMID 22117037
- [Background] Buxton AE. Implantable cardioverter-defibrillators for primary prevention of sudden death: the quest to identify patients most likely to benefit. J Am Coll Cardiol. 2012 Oct 23;60(17):1656-8. doi: 10.1016/j.jacc.2012.06.041. Epub 2012 Sep 26. No abstract available. PMID 23021332
- [Derived] Pelli A, Junttila MJ, Kentta TV, Schlogl S, Zabel M, Malik M, Reichlin T, Willems R, Vos MA, Harden M, Friede T, Sticherling C, Huikuri HV; EU-CERT-ICD Study Investigators. Q waves are the strongest electrocardiographic variable associated with primary prophylactic implantable cardioverter-defibrillator benefit: a prospective multicentre study. Europace. 2022 May 3;24(5):774-783. doi: 10.1093/europace/euab260. PMID 34849744
- [Derived] Dornquast C, Dombrowski M, Zabel M, Willich SN, Reinhold T. Potential drug-drug interactions in patients with indication for prophylactic implantation of a cardioverter defibrillator: a cross-sectional analysis. BMC Health Serv Res. 2020 Mar 31;20(1):271. doi: 10.1186/s12913-020-05131-7. PMID 32234046
- [Derived] Junttila MJ, Pelli A, Kentta TV, Friede T, Willems R, Bergau L, Malik M, Vandenberk B, Vos MA, Schmidt G, Merkely B, Lubinski A, Svetlosak M, Braunschweig F, Harden M, Zabel M, Huikuri HV, Sticherling C; EU-CERT-ICD Investigators. Appropriate Shocks and Mortality in Patients With Versus Without Diabetes With Prophylactic Implantable Cardioverter Defibrillators. Diabetes Care. 2020 Jan;43(1):196-200. doi: 10.2337/dc19-1014. Epub 2019 Oct 23. PMID 31645407
- See also: EU-CERT-ICD Website — http://www.eu-cert-icd.eu